CLINICAL TRIAL: NCT02120833
Title: A Multi-Center Clinical Trial to Evaluate the Efficacy of an Over-the-Counter Cream in the Management of Mild to Moderate Atopic Dermatitis in Infants and Toddlers
Brief Title: A Test to Determine the Usefulness and Safety of a Cream Used on Babies With Dry Itchy Skin
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CO-140206110636-SBCT
Record Dates: First submitted 2014-03-28; First posted 2014-04-23 (Estimated); Results first posted 2015-09-07 (Estimated); Last update posted 2017-01-13 (Estimated); Status verified 2017-01

CONDITIONS: Eczema
Keywords: Atopic Dermatitis
MeSH Terms: conditions — Eczema; Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- EPI (Active Comparator)
  Interventions: Device: EpiCeram® Skin Barrier Emulsion
- NEE (Experimental)
  Interventions: Drug: Colloidal Oatmeal Cream

INTERVENTIONS:
Device: EpiCeram® Skin Barrier Emulsion — Device (including sham) Apply in a thin layer to the affected skin areas 2 times per day (or as needed) and massage gently into the skin as directed.
  Arms: EPI
Drug: Colloidal Oatmeal Cream — Drug (including placebo) Apply in a thin layer to the affected skin areas 2 times per day (or as needed) and massage gently into the skin as directed.
  Arms: NEE

SUMMARY:
This study is for infants with mild to moderate dry and itchy skin. This study will involve going to the doctor for 6 visits over 2 weeks. All participants' skin will be examined by a dermatologist to determine if they have atopic dermatitis and have an active mild to moderate eczema wound. Participant's parents/guardians will be asked a few questions to determine if their child qualifies for the study.

Then all participants' caregivers will complete a questionnaire at the beginning of the study. The child's skin will be examined to rate the level of their eczema and a trained examiner will grade the looks and symptoms of their eczema. All parents or guardians will be instructed how to apply the test product and how to record usage on a diary card and then apply the test product. The test product will be applied at least 2 times per day or more as needed on all body areas, including the face affected throughout the study.

One digital picture will be taken of one eczema wound. Another digital picture will be taken of the area around this wound. These pictures will be taken on Day 0 (Baseline), Day 3, and Day 14.

Once product is applied the skin will be examined for any adverse events and all participants' caregivers will complete a questionnaire on study day 1, 3, 7 and 14.

DETAILED DESCRIPTION:
This is a multi-center, two-arm clinical trial in participants aged 2 - 35 months with mild to moderate Atopic Dermatitis (AD) as determined by the study physician. A sufficient number of participants will be enrolled in this study to yield 40 participants who complete the trial, 30 in the investigational product group and 10 in the active control group.

The investigational and control (EpiCeram®) products will be used topically. Participant caregivers will be instructed to gently massage the assigned product into the participant's skin. The treatments will be applied at least 2 times per day on all body areas, including areas of the body and face affected by AD. No product should be applied within 4 hours of a site visit. These treatments will be used in place of the participant's current moisturizers and/or emollients.

Diaries will be completed by the participants' caregivers each day, beginning upon initiation of therapy and continuing until trial completion/discontinuation, and will include information on product application and use of rescue medication.

All participants will visit the clinical site for assessments at baseline (Day 0) and on Days 1, 2, 3, 7 and 14. Clinical assessments include the Eczema Area and Severity index (EASI) and Investigator's Global Atopic Dermatitis Assessment (IGADA). Instrumental assessment of hydration will be done using a Corneometer (Courage & Khazaka, Germany). Caregivers will also complete a questionnaire to assess product experience. The final visit will occur on Day 14 or on the day of participant withdrawal from the trial.

ELIGIBILITY:
Inclusion Criteria

1. Able to comprehend and follow the requirements of the study (including availability on scheduled visit dates) based upon research site personnel's assessment;
2. Caregiver is able and willing to provide written informed consent for the participant to participate in the trial;
3. Male or female of any race or ethnicity, 2 months to 35 months of age;
4. Diagnosed as having Atopic Dermatitis (AD) on the basis of the criteria defined by Hanifin and Rajka
5. Rated as having mild to moderate AD (graded between 3.0 and 7.5 inclusive) as per Rajka-Langeland severity index
6. Willing to stop all emollients, moisturizers and/or other skin barrier cream or emulsion treatments for the AD condition during the test period. If using corticosteroids (not Class I, II, or III) or immunomodulators at study entry, must be on a stable dose for a minimum of 1 month;
7. Willing to undergo a washout period of 2 days before the trial initiation where no use of moisturizers or emollients will be allowed; and
8. Willing and able to comply with scheduled visits, treatment plan, and other trial procedures.

Exclusion Criteria:

1. Known sensitivity to any investigational product ingredient;
2. Use of a therapeutic (over the counter or prescription) body wash that contains an active ingredient for eczema;
3. Participation in any clinical study within 30 days of Visit 1;
4. Relative, partner or staff of any clinical research site personnel;
5. Active infection of any type at the start of the study;
6. Severe AD as determined by the Rajka-Langeland Severity Index
7. AD requiring systemic, super-potent (Class I) or potent (Class II or III) topical corticosteroids. If a participant requires any of these medications as rescue therapy during the study, the participant will be discontinued from the trial;
8. Requires any inhaled or intranasal corticosteroids;
9. Other medical condition that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the participant inappropriate for entry into this study.

Ages: 2 Months to 35 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 51 (Actual)
Dates: Start 2014-03; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Nunez, Study Director — Johnson & Johnson Consumer and Personal Products Worldwide
Locations (2):
- United States (2):
  - Thomas J. Stephens and Associates, Colorado Research Center, Colorado Springs, Colorado
  - Thomas J. Stephens and Associates, Dallas Research Center, Richardson, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- 1% Colloidal Oatmeal Eczema Cream: 1% Colloidal Oatmeal Eczema Cream, thin layer twice a day
- EpiCeram® Skin Barrier Emulsion: EpiCeram® Skin Barrier Emulsion, thin layer twice a day
Period: Overall Study
Arm/Group | 1% Colloidal Oatmeal Eczema Cream | EpiCeram® Skin Barrier Emulsion
Started | 39 | 12
Completed | 35 | 11
Not Completed | 4 | 1
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1% Colloidal Oatmeal Eczema Cream | EpiCeram® Skin Barrier Emulsion | Total
Number analyzed (Participants) | 39 | 12 | 51
Age, Continuous [Mean (Standard Deviation); unit: months] | 19.4 (9.78) | 22.3 (10.29) | 20.1 (9.88)
Gender [Count of Participants; unit: Participants]
  Female | 22 | 3 | 25
  Male | 17 | 9 | 26
Region of Enrollment [Number; unit: participants]
  USA | 39 | 12 | 51

OUTCOME MEASURES:

1. Primary Outcome: Eczema Area and Severity Index (EASI) on Day 3 - Change From Baseline
Description: The surface and severity of eczema is measured using the Eczema Area and Severity Index (EASI). A regional body surface area tabulation based on severity ranging from 0 (none) to 3 (severe), and severity of signs of disease, then multiplied by body area with final calculation ranging from 0-72.
Time Frame: Baseline to Day 3
Population: Analysis was based on Intent-to-Treat subjects, which included all randomized subjects.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1% Colloidal Oatmeal Eczema Cream | EpiCeram® Skin Barrier Emulsion
Number analyzed (Participants) | 30 | 9
units on a scale | -1.783 (1.72) | -0.767 (2.08)
Statistical Analysis 1: Comparison: 1% Colloidal Oatmeal Eczema Cream; The null hypothesis was no difference versus baseline. The alternative hypothesis was a difference versus baseline; Test type: Superiority or Other; p < 0.0001, One-sample t-test — The significance level threshold level was 0.05 (two-sided); Adjusted by study site
Statistical Analysis 2: Comparison: EpiCeram® Skin Barrier Emulsion; The null hypothesis was no difference versus baseline. The alternative hypothesis was a difference versus baseline; Test type: Superiority or Other; p = 0.4360, One-sample t-test — The significance level threshold level was 0.05 (two-sided); Adjusted by study site
Statistical Analysis 3: Comparison: 1% Colloidal Oatmeal Eczema Cream vs EpiCeram® Skin Barrier Emulsion; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.0510, ANCOVA — The significance threshold level was 0.05 (two-sided); Treatment and study site as factors, baseline score as covariate; Mean Difference (Final Values) = -1.25, 95% CI 2-sided [-2.51 to 0.01], Standard Error of Mean 0.62

2. Primary Outcome: Investigator's Global Atopic Dermatitis Assessment (IGADA) on Day 3 - Change From Baseline
Description: The signs and symptoms of eczema are measured using the Investigator's Global Atopic Dermatitis Assessment (IGADA). An assessment of atopic dermatitis based on a 4 point scale, ranging from 0 (none) and 3 (severe), is used to describe signs and symptoms in 4 designated body regions. Based on the presence or absence of the total number of signs and symptoms, the final rating is categorized as clear, almost clear, mild, moderate, severe, or very severe.
Time Frame: Baseline to Day 3
Population: Analysis was based on Intent-to-Treat subjects, which included all randomized subjects.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1% Colloidal Oatmeal Eczema Cream | EpiCeram® Skin Barrier Emulsion
Number analyzed (Participants) | 34 | 11
units on a scale | -0.441 (0.66) | -0.364 (0.50)
Statistical Analysis 1: Comparison: 1% Colloidal Oatmeal Eczema Cream; The null hypothesis was no difference versus baseline. The alternative hypothesis was a difference versus baseline; Test type: Superiority or Other; p = 0.0004, One-sample t-test — The significance level threshold level was 0.05 (two-sided); Adjusted by study site
Statistical Analysis 2: Comparison: EpiCeram® Skin Barrier Emulsion; The null hypothesis was no difference versus baseline. The alternative hypothesis was a difference versus baseline; Test type: Superiority or Other; p = 0.0213, One-sample t-test — The significance level threshold level was 0.05 (two-sided); Adjusted by study site
Statistical Analysis 3: Comparison: 1% Colloidal Oatmeal Eczema Cream vs EpiCeram® Skin Barrier Emulsion; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.7698, ANCOVA; The significance threshold level was 0.05 (two-sided); Mean Difference (Final Values) = -0.06, 95% CI 2-sided [-0.50 to 0.37], Standard Error of Mean 0.22

3. Secondary Outcome: Eczema Area and Severity Index (EASI) on Day 1 - Change From Baseline
Description: as for outcome 1
Time Frame: Baseline to Day 1
Population: Analysis was based on Intent-to-Treat subjects, which included all randomized subjects.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1% Colloidal Oatmeal Eczema Cream | EpiCeram® Skin Barrier Emulsion
Number analyzed (Participants) | 32 | 8
units on a scale | -0.672 (0.92) | -0.438 (1.65)
Statistical Analysis 1: Comparison: 1% Colloidal Oatmeal Eczema Cream; The null hypothesis was no difference versus baseline. The alternative hypothesis was a difference versus baseline; Test type: Superiority or Other; p = 0.0003, One-sample t-test — The significance level threshold level was 0.05 (two-sided); Adjusted by study site
Statistical Analysis 2: Comparison: EpiCeram® Skin Barrier Emulsion; The null hypothesis was no difference versus baseline. The alternative hypothesis was a difference versus baseline; Test type: Superiority or Other; p = 0.6063, One-sample t-test — The significance level threshold level was 0.05 (two-sided); Adjusted by study site
Statistical Analysis 3: Comparison: 1% Colloidal Oatmeal Eczema Cream vs EpiCeram® Skin Barrier Emulsion; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.3686, ANCOVA — The significance threshold level was 0.05 (two-sided); Treatment and study site as factors, baseline score as covariate; Mean Difference (Final Values) = -0.39, 95% CI 2-sided [-1.27 to 0.48], Standard Error of Mean 0.43

4. Secondary Outcome: Eczema Area and Severity Index (EASI) on Day 2 - Change From Baseline
Description: as for outcome 1
Time Frame: Baseline to Day 2
Population: Analysis was based on Intent-to-Treat subjects, which included all randomized subjects.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1% Colloidal Oatmeal Eczema Cream | EpiCeram® Skin Barrier Emulsion
Number analyzed (Participants) | 31 | 9
units on a scale | -1.194 (1.10) | -0.489 (2.49)
Statistical Analysis 1: Comparison: 1% Colloidal Oatmeal Eczema Cream; The null hypothesis was no difference versus baseline. The alternative hypothesis was a difference versus baseline; Test type: Superiority or Other; p < 0.0001, One-sample t-test — The significance level threshold level was 0.05 (two-sided); Adjusted by study site
Statistical Analysis 2: Comparison: EpiCeram® Skin Barrier Emulsion; The null hypothesis was no difference versus baseline. The alternative hypothesis was a difference versus baseline; Test type: Superiority or Other; p = 0.6118, One-sample t-test — The significance level threshold level was 0.05 (two-sided); Adjusted by study site
Statistical Analysis 3: Comparison: 1% Colloidal Oatmeal Eczema Cream vs EpiCeram® Skin Barrier Emulsion; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.1485, ANCOVA — The significance threshold level was 0.05 (two-sided); Treatment and study site as factors, baseline score as covariate; Mean Difference (Final Values) = -0.83, 95% CI 2-sided [-1.98 to 0.31], Standard Error of Mean 0.56

5. Secondary Outcome: Eczema Area and Severity Index (EASI) on Day 7 - Change From Baseline
Description: as for outcome 1
Time Frame: Baseline to Day 7
Population: Analysis was based on Intent-to-Treat subjects, which included all randomized subjects.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1% Colloidal Oatmeal Eczema Cream | EpiCeram® Skin Barrier Emulsion
Number analyzed (Participants) | 30 | 9
units on a scale | -2.410 (2.49) | -1.233 (1.41)
Statistical Analysis 1: Comparison: 1% Colloidal Oatmeal Eczema Cream; The null hypothesis was no difference versus baseline. The alternative hypothesis was a difference versus baseline; Test type: Superiority or Other; p < 0.0001, One-sample t-test — The significance level threshold level was 0.05 (two-sided); Adjusted by study site
Statistical Analysis 2: Comparison: EpiCeram® Skin Barrier Emulsion; The null hypothesis was no difference versus baseline. The alternative hypothesis was a difference versus baseline; Test type: Superiority or Other; p = 0.2447, One-sample t-test — The significance level threshold level was 0.05 (two-sided); Adjusted by study site
Statistical Analysis 3: Comparison: 1% Colloidal Oatmeal Eczema Cream vs EpiCeram® Skin Barrier Emulsion; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.0216, ANCOVA — The significance threshold level was 0.05 (two-sided); Treatment and study site as factors, baseline score as covariate; Mean Difference (Final Values) = -1.60, 95% CI 2-sided [-2.95 to -0.25], Standard Error of Mean 0.67

6. Secondary Outcome: Eczema Area and Severity Index (EASI) on Day 14 - Change From Baseline
Description: as for outcome 1
Time Frame: Baseline to Day 14
Population: Analysis was based on Intent-to-Treat subjects, which included all randomized subjects.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1% Colloidal Oatmeal Eczema Cream | EpiCeram® Skin Barrier Emulsion
Number analyzed (Participants) | 31 | 9
units on a scale | -2.403 (2.30) | -1.833 (2.74)
Statistical Analysis 1: Comparison: 1% Colloidal Oatmeal Eczema Cream; The null hypothesis was no difference versus baseline. The alternative hypothesis was a difference versus baseline; Test type: Superiority or Other; p < 0.0001, One-sample t-test — The significance level threshold level was 0.05 (two-sided); Adjusted by study site
Statistical Analysis 2: Comparison: EpiCeram® Skin Barrier Emulsion; The null hypothesis was no difference versus baseline. The alternative hypothesis was a difference versus baseline; Test type: Superiority or Other; p = 0.0476, One-sample t-test — The significance level threshold level was 0.05 (two-sided); Adjusted by study site
Statistical Analysis 3: Comparison: 1% Colloidal Oatmeal Eczema Cream vs EpiCeram® Skin Barrier Emulsion; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.2349, ANCOVA — The significance threshold level was 0.05 (two-sided); Treatment and study site as factors, baseline score as covariate; Mean Difference (Final Values) = -0.94, 95% CI 2-sided [-2.52 to 0.64], Standard Error of Mean 0.78

7. Secondary Outcome: Investigator's Global Atopic Dermatitis Assessment (IGADA) on Day 1 - Change From Baseline
Description: as for outcome 2
Time Frame: Baseline to Day 1
Population: Analysis was based on Intent-to-Treat subjects, which included all randomized subjects.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1% Colloidal Oatmeal Eczema Cream | EpiCeram® Skin Barrier Emulsion
Number analyzed (Participants) | 37 | 10
units on a scale | -0.027 (0.16) | -0.100 (0.32)
Statistical Analysis 1: Comparison: 1% Colloidal Oatmeal Eczema Cream; The null hypothesis was no difference versus baseline. The alternative hypothesis was a difference versus baseline; Test type: Superiority or Other; p = 0.7842, One-sample t-test — The significance level threshold level was 0.05 (two-sided); Adjusted by study site
Statistical Analysis 2: Comparison: EpiCeram® Skin Barrier Emulsion; The null hypothesis was no difference versus baseline. The alternative hypothesis was a difference versus baseline; Test type: Superiority or Other; p = 0.6083, One-sample t-test — The significance level threshold level was 0.05 (two-sided); Adjusted by study site
Statistical Analysis 3: Comparison: 1% Colloidal Oatmeal Eczema Cream vs EpiCeram® Skin Barrier Emulsion; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.3599, ANCOVA — The significance threshold level was 0.05 (two-sided); Treatment and study site as factors, baseline score as covariate; Mean Difference (Final Values) = 0.07, 95% CI 2-sided [-0.08 to 0.22], Standard Error of Mean 0.07

8. Secondary Outcome: Investigator's Global Atopic Dermatitis Assessment (IGADA) on Day 2 - Change From Baseline
Description: as for outcome 2
Time Frame: Baseline to Day 2
Population: Analysis was based on Intent-to-Treat subjects, which included all randomized subjects.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1% Colloidal Oatmeal Eczema Cream | EpiCeram® Skin Barrier Emulsion
Number analyzed (Participants) | 36 | 11
units on a scale | -0.417 (0.55) | -0.364 (0.50)
Statistical Analysis 1: Comparison: 1% Colloidal Oatmeal Eczema Cream; The null hypothesis was no difference versus baseline. The alternative hypothesis was a difference versus baseline; Test type: Superiority or Other; p = 0.0001, One-sample t-test — The significance level threshold level was 0.05 (two-sided); Adjusted by study site
Statistical Analysis 2: Comparison: EpiCeram® Skin Barrier Emulsion; The null hypothesis was no difference versus baseline. The alternative hypothesis was a difference versus baseline; Test type: Superiority or Other; p = 0.0317, One-sample t-test — The significance level threshold level was 0.05 (two-sided); Adjusted by study site
Statistical Analysis 3: Comparison: 1% Colloidal Oatmeal Eczema Cream vs EpiCeram® Skin Barrier Emulsion; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.8037, ANCOVA — The significance threshold level was 0.05 (two-sided); Treatment and study site as factors, baseline score as covariate; Mean Difference (Final Values) = -0.05, 95% CI 2-sided [-0.42 to 0.33], Standard Error of Mean 0.19

9. Secondary Outcome: Investigator's Global Atopic Dermatitis Assessment (IGADA) on Day 7 - Change From Baseline
Description: as for outcome 2
Time Frame: Baseline to Day 7
Population: Analysis was based on Intent-to-Treat subjects, which included all randomized subjects.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1% Colloidal Oatmeal Eczema Cream | EpiCeram® Skin Barrier Emulsion
Number analyzed (Participants) | 35 | 11
units on a scale | -0.743 (0.66) | -0.364 (0.50)
Statistical Analysis 1: Comparison: 1% Colloidal Oatmeal Eczema Cream; The null hypothesis was no difference versus baseline. The alternative hypothesis was a difference versus baseline; Test type: Superiority or Other; p < 0.0001, One-sample t-test — The significance level threshold level was 0.05 (two-sided); Adjusted by study site
Statistical Analysis 2: Comparison: EpiCeram® Skin Barrier Emulsion; The null hypothesis was no difference versus baseline. The alternative hypothesis was a difference versus baseline; Test type: Superiority or Other; p = 0.0244, One-sample t-test — The significance level threshold level was 0.05 (two-sided); Adjusted by study site
Statistical Analysis 3: Comparison: 1% Colloidal Oatmeal Eczema Cream vs EpiCeram® Skin Barrier Emulsion; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.0900, ANCOVA — The significance threshold level was 0.05 (two-sided); Treatment and study site as factors, baseline score as covariate; Mean Difference (Final Values) = -0.37, 95% CI 2-sided [-0.80 to 0.06], Standard Error of Mean 0.21

10. Secondary Outcome: Investigator's Global Atopic Dermatitis Assessment (IGADA) on Day 14 - Change From Baseline
Description: as for outcome 2
Time Frame: Baseline to Day 14
Population: Analysis was based on Intent-to-Treat subjects, which included all randomized subjects.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1% Colloidal Oatmeal Eczema Cream | EpiCeram® Skin Barrier Emulsion
Number analyzed (Participants) | 36 | 11
units on a scale | -0.861 (0.90) | -0.455 (0.52)
Statistical Analysis 1: Comparison: 1% Colloidal Oatmeal Eczema Cream; The null hypothesis was no difference versus baseline. The alternative hypothesis was a difference versus baseline; Test type: Superiority or Other; p < 0.0001, One-sample t-test — The significance level threshold level was 0.05 (two-sided); Adjusted by study site
Statistical Analysis 2: Comparison: EpiCeram® Skin Barrier Emulsion; The null hypothesis was no difference versus baseline. The alternative hypothesis was a difference versus baseline; Test type: Superiority or Other; p = 0.0065, One-sample t-test — The significance level threshold level was 0.05 (two-sided); Adjusted by study site
Statistical Analysis 3: Comparison: 1% Colloidal Oatmeal Eczema Cream vs EpiCeram® Skin Barrier Emulsion; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.1561, ANCOVA — The significance threshold level was 0.05 (two-sided); Treatment and study site as factors, baseline score as covariate; Mean Difference (Final Values) = -0.40, 95% CI 2-sided [-0.97 to 0.16], Standard Error of Mean 0.28

11. Secondary Outcome: Corneometer Measurement on Day 0 - Post-Treatment - Change From Baseline
Description: Corneometer is a non-invasive instrument that measures hydration on the skin surface. During assessment, the corneometer was placed at a site adjacent to eczema-affected skin areas. Corneometer readings are directly related to the skin's electrical capacitance and increase as the skin becomes more hydrated. Pre-treatment readings ranged from 2.0 to 68.0. Post-treatment on Day 0, corneometer readings ranged from 10.3 to 86.3.
Time Frame: Baseline to Post -Treatment on Day 0
Population: Analysis was based on Intent-to-Treat subjects, which included all randomized subjects.
Measure: Mean (Standard Deviation); unit: arbitrary units
Arm/Group | 1% Colloidal Oatmeal Eczema Cream | EpiCeram® Skin Barrier Emulsion
Number analyzed (Participants) | 39 | 12
arbitrary units | 17.277 (14.58) | 11.544 (12.43)
Statistical Analysis 1: Comparison: 1% Colloidal Oatmeal Eczema Cream; The null hypothesis was no difference versus baseline. The alternative hypothesis was a difference versus baseline; Test type: Superiority or Other; p < 0.0001, One-sample t-test — The significance level threshold level was 0.05 (two-sided); Adjusted by study site
Statistical Analysis 2: Comparison: EpiCeram® Skin Barrier Emulsion; The null hypothesis was no difference versus baseline. The alternative hypothesis was a difference versus baseline; Test type: Superiority or Other; p = 0.0049, One-sample t-test — The significance level threshold level was 0.05 (two-sided); Adjusted by study site
Statistical Analysis 3: Comparison: 1% Colloidal Oatmeal Eczema Cream vs EpiCeram® Skin Barrier Emulsion; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.2409, ANCOVA — The significance threshold level was 0.05 (two-sided); Treatment and study site as factors, baseline score as covariate; Mean Difference (Final Values) = 5.59, 95% CI 2-sided [-3.88 to 15.07], Standard Error of Mean 4.71

12. Secondary Outcome: Corneometer Measurement on Day 1 - Change From Baseline
Description: Corneometer is a non-invasive instrument that measures hydration on the skin surface. During assessment, the corneometer was placed at a site adjacent to eczema-affected skin areas. Corneometer readings are directly related to the skin's electrical capacitance and increase as the skin becomes more hydrated. Pre-treatment readings ranged from 2.0 to 68.0. On Day 1, corneometer readings ranged from 5.5 to 84.0.
Time Frame: Baseline to Day 1
Population: Analysis was based on Intent-to-Treat subjects, which included all randomized subjects.
Measure: Mean (Standard Deviation); unit: arbitrary units
Arm/Group | 1% Colloidal Oatmeal Eczema Cream | EpiCeram® Skin Barrier Emulsion
Number analyzed (Participants) | 37 | 10
arbitrary units | 15.182 (11.57) | 6.483 (13.37)
Statistical Analysis 1: Comparison: 1% Colloidal Oatmeal Eczema Cream; The null hypothesis was no difference versus baseline. The alternative hypothesis was a difference versus baseline; Test type: Superiority or Other; p < 0.0001, One-sample t-test — The significance level threshold level was 0.05 (two-sided); Adjusted by study site
Statistical Analysis 2: Comparison: EpiCeram® Skin Barrier Emulsion; The null hypothesis was no difference versus baseline. The alternative hypothesis was a difference versus baseline; Test type: Superiority or Other; p = 0.2386, One-sample t-test — The significance level threshold level was 0.05 (two-sided); Adjusted by study site
Statistical Analysis 3: Comparison: 1% Colloidal Oatmeal Eczema Cream vs EpiCeram® Skin Barrier Emulsion; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.0241, ANCOVA — The significance threshold level was 0.05 (two-sided); Treatment and study site as factors, baseline score as covariate; Mean Difference (Final Values) = 9.30, 95% CI 2-sided [1.28 to 17.32], Standard Error of Mean 3.98

13. Secondary Outcome: Corneometer Measurement on Day 2 - Change From Baseline
Description: Corneometer is a non-invasive instrument that measures hydration on the skin surface. During assessment, the corneometer was placed at a site adjacent to eczema-affected skin areas. Corneometer readings are directly related to the skin's electrical capacitance and increase as the skin becomes more hydrated. Pre-treatment readings ranged from 2.0 to 68.0. On Day 2, corneometer readings ranged from 8.5 to 74.0.
Time Frame: Baseline to Day 2
Population: Analysis was based on Intent-to-Treat subjects, which included all randomized subjects.
Measure: Mean (Standard Deviation); unit: arbitrary units
Arm/Group | 1% Colloidal Oatmeal Eczema Cream | EpiCeram® Skin Barrier Emulsion
Number analyzed (Participants) | 36 | 11
arbitrary units | 17.019 (13.50) | 7.864 (10.96)
Statistical Analysis 1: Comparison: 1% Colloidal Oatmeal Eczema Cream; The null hypothesis was no difference versus baseline. The alternative hypothesis was a difference versus baseline; Test type: Superiority or Other; p < 0.0001, One-sample t-test — The significance level threshold level was 0.05 (two-sided); Adjusted by study site
Statistical Analysis 2: Comparison: EpiCeram® Skin Barrier Emulsion; The null hypothesis was no difference versus baseline. The alternative hypothesis was a difference versus baseline; Test type: Superiority or Other; p = 0.0696, One-sample t-test — The significance level threshold level was 0.05 (two-sided); Adjusted by study site
Statistical Analysis 3: Comparison: 1% Colloidal Oatmeal Eczema Cream vs EpiCeram® Skin Barrier Emulsion; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.0394, ANCOVA — The significance threshold level was 0.05 (two-sided); Treatment and study site as factors, baseline score as covariate; Mean Difference (Final Values) = 8.99, 95% CI 2-sided [0.46 to 17.52], Standard Error of Mean 4.23

14. Secondary Outcome: Corneometer Measurement on Day 3 - Change From Baseline
Description: Corneometer is a non-invasive instrument that measures hydration on the skin surface. During assessment, the corneometer was placed at a site adjacent to eczema-affected skin areas. Corneometer readings are directly related to the skin's electrical capacitance and increase as the skin becomes more hydrated. Pre-treatment readings ranged from 2.0 to 68.0. On Day 3, corneometer readings ranged from 8.0 to 65.3.
Time Frame: Baseline to Day 3
Population: Analysis was based on Intent-to-Treat subjects, which included all randomized subjects.
Measure: Mean (Standard Deviation); unit: arbitrary units
Arm/Group | 1% Colloidal Oatmeal Eczema Cream | EpiCeram® Skin Barrier Emulsion
Number analyzed (Participants) | 34 | 11
arbitrary units | 16.276 (11.61) | 7.661 (11.01)
Statistical Analysis 1: Comparison: 1% Colloidal Oatmeal Eczema Cream; The null hypothesis was no difference versus baseline. The alternative hypothesis was a difference versus baseline; Test type: Superiority or Other; p < 0.0001, One-sample t-test — The significance level threshold level was 0.05 (two-sided); Adjusted by study site
Statistical Analysis 2: Comparison: EpiCeram® Skin Barrier Emulsion; The null hypothesis was no difference versus baseline. The alternative hypothesis was a difference versus baseline; Test type: Superiority or Other; p = 0.0772, One-sample t-test — The significance level threshold level was 0.05 (two-sided); Adjusted by study site
Statistical Analysis 3: Comparison: 1% Colloidal Oatmeal Eczema Cream vs EpiCeram® Skin Barrier Emulsion; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.0213, ANCOVA — The significance threshold level was 0.05 (two-sided); Treatment and study site as factors, baseline score as covariate; Mean Difference (Final Values) = 8.48, 95% CI 2-sided [1.33 to 15.63], Standard Error of Mean 3.54

15. Secondary Outcome: Corneometer Measurement on Day 7 - Change From Baseline
Description: Corneometer is a non-invasive instrument that measures hydration on the skin surface. During assessment, the corneometer was placed at a site adjacent to eczema-affected skin areas. Corneometer readings are directly related to the skin's electrical capacitance and increase as the skin becomes more hydrated. Pre-treatment readings ranged from 2.0 to 68.0. On Day 7, corneometer readings ranged from 6.8 to 65.0.
Time Frame: Baseline to Day 7
Population: Analysis was based on Intent-to-Treat subjects, which included all randomized subjects.
Measure: Mean (Standard Deviation); unit: arbitrary units
Arm/Group | 1% Colloidal Oatmeal Eczema Cream | EpiCeram® Skin Barrier Emulsion
Number analyzed (Participants) | 35 | 11
arbitrary units | 15.167 (11.33) | 10.318 (16.01)
Statistical Analysis 1: Comparison: 1% Colloidal Oatmeal Eczema Cream; The null hypothesis was no difference versus baseline. The alternative hypothesis was a difference versus baseline; Test type: Superiority or Other; p < 0.0001, One-sample t-test — The significance level threshold level was 0.05 (two-sided); Adjusted by study site
Statistical Analysis 2: Comparison: EpiCeram® Skin Barrier Emulsion; The null hypothesis was no difference versus baseline. The alternative hypothesis was a difference versus baseline; Test type: Superiority or Other; p = 0.0172, One-sample t-test — The significance level threshold level was 0.05 (two-sided); Adjusted by study site
Statistical Analysis 3: Comparison: 1% Colloidal Oatmeal Eczema Cream vs EpiCeram® Skin Barrier Emulsion; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.1968, ANCOVA — The significance threshold level was 0.05 (two-sided); Treatment and study site as factors, baseline score as covariate; Mean Difference (Final Values) = 4.56, 95% CI 2-sided [-2.46 to 11.58], Standard Error of Mean 3.48

16. Secondary Outcome: Corneometer Measurement on Day 14 - Change From Baseline
Description: Corneometer is a non-invasive instrument that measures hydration on the skin surface. During assessment, the corneometer was placed at a site adjacent to eczema-affected skin areas. Corneometer readings are directly related to the skin's electrical capacitance and increase as the skin becomes more hydrated. Pre-treatment readings ranged from 2.0 to 68.0. On Day 14, corneometer readings ranged from 5.7 to 73.1.
Time Frame: Baseline to Day 14
Population: Analysis was based on Intent-to-Treat subjects, which included all randomized subjects.
Measure: Mean (Standard Deviation); unit: arbitrary units
Arm/Group | 1% Colloidal Oatmeal Eczema Cream | EpiCeram® Skin Barrier Emulsion
Number analyzed (Participants) | 36 | 11
arbitrary units | 15.253 (9.79) | 7.818 (12.58)
Statistical Analysis 1: Comparison: 1% Colloidal Oatmeal Eczema Cream; The null hypothesis was no difference versus baseline. The alternative hypothesis was a difference versus baseline; Test type: Superiority or Other; p < 0.0001, One-sample t-test — The significance level threshold level was 0.05 (two-sided); Adjusted by study site
Statistical Analysis 2: Comparison: EpiCeram® Skin Barrier Emulsion; The null hypothesis was no difference versus baseline. The alternative hypothesis was a difference versus baseline; Test type: Superiority or Other; p = 0.0712, One-sample t-test — The significance level threshold level was 0.05 (two-sided); Adjusted by study site
Statistical Analysis 3: Comparison: 1% Colloidal Oatmeal Eczema Cream vs EpiCeram® Skin Barrier Emulsion; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.0313, ANCOVA — The significance threshold level was 0.05 (two-sided); Treatment and study site as factors, baseline score as covariate; Mean Difference (Final Values) = 7.43, 95% CI 2-sided [0.70 to 14.15], Standard Error of Mean 3.34

17. Secondary Outcome: Caregiver Questionnaire on Day 0 Pre-treatment - Overall, my Baby's Skin Looks Smooth
Description: Questions were answered before treatment by participant's caregiver. Questions included overall look (smooth, healthy) and feel (soft, smooth) of participant's skin, and affected area's look (smooth, healthy) and feel (soft, smooth). Caregiver answered based on a 6 point system from 'I don't have an opinion' to 'strongly disagree.'
Time Frame: 0 Days - Pre-Treatment
Population: Analysis was based on Intent-to-Treat subjects, which included all randomized subjects.
Measure: Number; unit: participants
Arm/Group | 1% Colloidal Oatmeal Eczema Cream | EpiCeram® Skin Barrier Emulsion
Number analyzed (Participants) | 39 | 12
participants
  I don't have an opinion | 0 | 0
  Strongly disagree | 9 | 2
  Somewhat disagree | 12 | 2
  Neither agree nor disagree | 3 | 1
  Somewhat agree | 13 | 5
  Strongly agree | 2 | 2
  Missing | 0 | 0

18. Secondary Outcome: Caregiver Questionnaire on Day 0 Pre-treatment - Overall, my Baby's Skin Looks Healthy
Description: as for outcome 17
Time Frame: 0 Days - Pre-Treatment
Population: Analysis was based on Intent-to-Treat subjects, which included all randomized subjects.
Measure: Number; unit: participants
Arm/Group | 1% Colloidal Oatmeal Eczema Cream | EpiCeram® Skin Barrier Emulsion
Number analyzed (Participants) | 39 | 12
participants
  I don't have an opinion | 0 | 0
  Strongly disagree | 0 | 1
  Somewhat disagree | 17 | 4
  Neither agree nor disagree | 5 | 1
  Somewhat agree | 12 | 4
  Strongly agree | 5 | 2
  Missing | 0 | 0

19. Secondary Outcome: Caregiver Questionnaire on Day 0 Pre-treatment - Overall, my Baby's Skin Feels Soft
Description: as for outcome 17
Time Frame: 0 Days - Pre-Treatment
Population: Analysis was based on Intent-to-Treat subjects, which included all randomized subjects.
Measure: Number; unit: participants
Arm/Group | 1% Colloidal Oatmeal Eczema Cream | EpiCeram® Skin Barrier Emulsion
Number analyzed (Participants) | 39 | 12
participants
  I don't have an opinion | 0 | 0
  Strongly disagree | 5 | 2
  Somewhat disagree | 13 | 3
  Neither agree nor disagree | 4 | 1
  Somewhat agree | 14 | 4
  Strongly agree | 3 | 2
  Missing | 0 | 0

20. Secondary Outcome: Caregiver Questionnaire on Day 0 Pre-treatment - Overall, my Baby's Skin Feels Smooth
Description: as for outcome 17
Time Frame: 0 Days - Pre-Treatment
Population: Analysis was based on Intent-to-Treat subjects, which included all randomized subjects.
Measure: Number; unit: participants
Arm/Group | 1% Colloidal Oatmeal Eczema Cream | EpiCeram® Skin Barrier Emulsion
Number analyzed (Participants) | 39 | 12
participants
  I don't have an opinion | 0 | 0
  Strongly disagree | 6 | 2
  Somewhat disagree | 13 | 5
  Neither agree nor disagree | 4 | 1
  Somewhat agree | 13 | 2
  Strongly agree | 2 | 2
  Missing | 1 | 0

21. Secondary Outcome: Caregiver Questionnaire on Day 0 Pre-treatment - In the Areas Affected by Eczema, my Baby's Skin Looks Smooth
Description: as for outcome 17
Time Frame: 0 Days - Pre-Treatment
Population: Analysis was based on Intent-to-Treat subjects, which included all randomized subjects.
Measure: Number; unit: participants
Arm/Group | 1% Colloidal Oatmeal Eczema Cream | EpiCeram® Skin Barrier Emulsion
Number analyzed (Participants) | 39 | 12
participants
  I don't have an opinion | 0 | 0
  Strongly disagree | 22 | 8
  Somewhat disagree | 12 | 4
  Neither agree nor disagree | 1 | 0
  Somewhat agree | 4 | 0
  Strongly agree | 0 | 0
  Missing | 0 | 0

22. Secondary Outcome: Caregiver Questionnaire on Day 0 Pre-treatment - In the Areas Affected by Eczema, my Baby's Skin Looks Healthy
Description: as for outcome 17
Time Frame: 0 Days - Pre-Treatment
Population: Analysis was based on Intent-to-Treat subjects, which included all randomized subjects.
Measure: Number; unit: participants
Arm/Group | 1% Colloidal Oatmeal Eczema Cream | EpiCeram® Skin Barrier Emulsion
Number analyzed (Participants) | 39 | 12
participants
  I don't have an opinion | 0 | 0
  Strongly disagree | 17 | 4
  Somewhat disagree | 15 | 8
  Neither agree nor disagree | 3 | 0
  Somewhat agree | 4 | 0
  Strongly agree | 0 | 0
  Missing | 0 | 0

23. Secondary Outcome: Caregiver Questionnaire on Day 0 Pre-treatment - In the Areas Affected by Eczema, my Baby's Skin Feels Soft
Description: as for outcome 17
Time Frame: 0 Days - Pre-Treatment
Population: Analysis was based on Intent-to-Treat subjects, which included all randomized subjects.
Measure: Number; unit: participants
Arm/Group | 1% Colloidal Oatmeal Eczema Cream | EpiCeram® Skin Barrier Emulsion
Number analyzed (Participants) | 39 | 12
participants
  I don't have an opinion | 0 | 0
  Strongly disagree | 21 | 8
  Somewhat disagree | 10 | 4
  Neither agree nor disagree | 3 | 0
  Somewhat agree | 4 | 0
  Strongly agree | 1 | 0
  Missing | 0 | 0

24. Secondary Outcome: Caregiver Questionnaire on Day 0 Pre-treatment - In the Areas Affected by Eczema, my Baby's Skin Feels Smooth
Description: as for outcome 17
Time Frame: 0 Days - Pre-Treatment
Population: Analysis was based on Intent-to-Treat subjects, which included all randomized subjects.
Measure: Number; unit: participants
Arm/Group | 1% Colloidal Oatmeal Eczema Cream | EpiCeram® Skin Barrier Emulsion
Number analyzed (Participants) | 39 | 12
participants
  I don't have an opinion | 0 | 0
  Strongly disagree | 21 | 8
  Somewhat disagree | 13 | 4
  Neither agree nor disagree | 0 | 0
  Somewhat agree | 5 | 0
  Strongly agree | 0 | 0
  Missing | 0 | 0

25. Secondary Outcome: Caregiver Questionnaire on Day 0 Post-treatment - Overall, my Baby's Skin Looks Smooth
Description: Questions were answered immediately post-treatment by participant's caregiver. Questions included overall look (smooth, healthy) and feel (soft, smooth) of participant's skin, and affected area's look (smooth, healthy) and feel (soft, smooth). Caregiver answered based on a 6 point system from 'I don't have an opinion' to 'strongly disagree.'
Time Frame: 0 Days - Post-Treatment
Population: Analysis was based on Intent-to-Treat subjects, which included all randomized subjects.
Measure: Number; unit: participants
Arm/Group | 1% Colloidal Oatmeal Eczema Cream | EpiCeram® Skin Barrier Emulsion
Number analyzed (Participants) | 39 | 12
participants
  I don't have an opinion | 0 | 0
  Strongly disagree | 2 | 1
  Somewhat disagree | 11 | 2
  Neither agree nor disagree | 4 | 3
  Somewhat agree | 14 | 4
  Strongly agree | 8 | 2
  Missing | 0 | 0

26. Secondary Outcome: Caregiver Questionnaire on Day 0 Post-treatment - Overall, my Baby's Skin Looks Healthy
Description: as for outcome 25
Time Frame: 0 Days - Post-Treatment
Population: Analysis was based on Intent-to-Treat subjects, which included all randomized subjects.
Measure: Number; unit: participants
Arm/Group | 1% Colloidal Oatmeal Eczema Cream | EpiCeram® Skin Barrier Emulsion
Number analyzed (Participants) | 39 | 12
participants
  I don't have an opinion | 0 | 0
  Strongly disagree | 1 | 1
  Somewhat disagree | 11 | 3
  Neither agree nor disagree | 4 | 1
  Somewhat agree | 19 | 5
  Strongly agree | 4 | 2
  Missing | 0 | 0

27. Secondary Outcome: Caregiver Questionnaire on Day 0 Post-treatment - Overall, my Baby's Skin Feels Soft
Description: as for outcome 25
Time Frame: 0 Days - Post-Treatment
Population: Analysis was based on Intent-to-Treat subjects, which included all randomized subjects.
Measure: Number; unit: participants
Arm/Group | 1% Colloidal Oatmeal Eczema Cream | EpiCeram® Skin Barrier Emulsion
Number analyzed (Participants) | 39 | 12
participants
  I don't have an opinion | 0 | 0
  Strongly disagree | 2 | 1
  Somewhat disagree | 10 | 2
  Neither agree nor disagree | 3 | 3
  Somewhat agree | 15 | 4
  Strongly agree | 9 | 2
  Missing | 0 | 0

28. Secondary Outcome: Caregiver Questionnaire on Day 0 Post-treatment - Overall, my Baby's Skin Feels Smooth
Description: as for outcome 25
Time Frame: 0 Days - Post-Treatment
Population: Analysis was based on Intent-to-Treat subjects, which included all randomized subjects.
Measure: Number; unit: participants
Arm/Group | 1% Colloidal Oatmeal Eczema Cream | EpiCeram® Skin Barrier Emulsion
Number analyzed (Participants) | 39 | 12
participants
  I don't have an opinion | 0 | 0
  Strongly disagree | 3 | 1
  Somewhat disagree | 7 | 3
  Neither agree nor disagree | 4 | 3
  Somewhat agree | 18 | 3
  Strongly agree | 7 | 2
  Missing | 0 | 0

29. Secondary Outcome: Caregiver Questionnaire on Day 0 Post-treatment - Overall, my Baby's Skin Feels Soft and Smooth Instantly
Description: as for outcome 25
Time Frame: 0 Days - Post-Treatment
Population: Analysis was based on Intent-to-Treat subjects, which included all randomized subjects.
Measure: Number; unit: participants
Arm/Group | 1% Colloidal Oatmeal Eczema Cream | EpiCeram® Skin Barrier Emulsion
Number analyzed (Participants) | 39 | 12
participants
  I don't have an opinion | 0 | 0
  Strongly disagree | 2 | 1
  Somewhat disagree | 5 | 2
  Neither agree nor disagree | 7 | 4
  Somewhat agree | 17 | 3
  Strongly agree | 8 | 2
  Missing | 0 | 0

30. Secondary Outcome: Caregiver Questionnaire on Day 0 Post-treatment - In the Areas Affected by Eczema, my Baby's Skin Looks Smooth
Description: as for outcome 25
Time Frame: 0 Days - Post-Treatment
Population: Analysis was based on Intent-to-Treat subjects, which included all randomized subjects.
Measure: Number; unit: participants
Arm/Group | 1% Colloidal Oatmeal Eczema Cream | EpiCeram® Skin Barrier Emulsion
Number analyzed (Participants) | 39 | 12
participants
  I don't have an opinion | 0 | 0
  Strongly disagree | 9 | 3
  Somewhat disagree | 9 | 3
  Neither agree nor disagree | 4 | 4
  Somewhat agree | 15 | 2
  Strongly agree | 2 | 0
  Missing | 0 | 0

31. Secondary Outcome: Caregiver Questionnaire on Day 0 Post-treatment - In the Areas Affected by Eczema, my Baby's Skin Looks Healthy
Description: as for outcome 25
Time Frame: 0 Days - Post-Treatment
Population: Analysis was based on Intent-to-Treat subjects, which included all randomized subjects.
Measure: Number; unit: participants
Arm/Group | 1% Colloidal Oatmeal Eczema Cream | EpiCeram® Skin Barrier Emulsion
Number analyzed (Participants) | 39 | 12
participants
  I don't have an opinion | 0 | 0
  Strongly disagree | 8 | 1
  Somewhat disagree | 9 | 8
  Neither agree nor disagree | 8 | 2
  Somewhat agree | 11 | 1
  Strongly agree | 3 | 0
  Missing | 0 | 0

32. Secondary Outcome: Caregiver Questionnaire on Day 0 Post-treatment - In the Areas Affected by Eczema, my Baby's Skin Feels Soft
Description: as for outcome 25
Time Frame: 0 Days - Post-Treatment
Population: Analysis was based on Intent-to-Treat subjects, which included all randomized subjects.
Measure: Number; unit: participants
Arm/Group | 1% Colloidal Oatmeal Eczema Cream | EpiCeram® Skin Barrier Emulsion
Number analyzed (Participants) | 39 | 12
participants
  I don't have an opinion | 0 | 0
  Strongly disagree | 8 | 2
  Somewhat disagree | 7 | 6
  Neither agree nor disagree | 4 | 1
  Somewhat agree | 13 | 3
  Strongly agree | 7 | 0
  Missing | 0 | 0

33. Secondary Outcome: Caregiver Questionnaire on Day 0 Post-treatment - In the Areas Affected by Eczema, my Baby's Skin Feels Smooth
Description: as for outcome 25
Time Frame: 0 Days - Post-Treatment
Population: Analysis was based on Intent-to-Treat subjects, which included all randomized subjects.
Measure: Number; unit: participants
Arm/Group | 1% Colloidal Oatmeal Eczema Cream | EpiCeram® Skin Barrier Emulsion
Number analyzed (Participants) | 39 | 12
participants
  I don't have an opinion | 0 | 0
  Strongly disagree | 7 | 2
  Somewhat disagree | 9 | 6
  Neither agree nor disagree | 3 | 1
  Somewhat agree | 12 | 3
  Strongly agree | 8 | 0
  Missing | 0 | 0

34. Secondary Outcome: Caregiver Questionnaire on Day 0 Post-treatment - In the Areas Affected by Eczema, my Baby's Skin Feels Soft and Smooth Instantly
Description: as for outcome 25
Time Frame: 0 Days - Post-Treatment
Population: Analysis was based on Intent-to-Treat subjects, which included all randomized subjects.
Measure: Number; unit: participants
Arm/Group | 1% Colloidal Oatmeal Eczema Cream | EpiCeram® Skin Barrier Emulsion
Number analyzed (Participants) | 39 | 12
participants
  I don't have an opinion | 0 | 0
  Strongly disagree | 6 | 1
  Somewhat disagree | 7 | 4
  Neither agree nor disagree | 6 | 4
  Somewhat agree | 10 | 3
  Strongly agree | 10 | 0
  Missing | 0 | 0

35. Secondary Outcome: Caregiver Questionnaire on Day 1 - Overall, my Baby's Skin Looks Smooth
Description: as for outcome 25
Time Frame: 1 Day
Population: Analysis was based on Intent-to-Treat subjects, which included all randomized subjects.
Measure: Number; unit: participants
Arm/Group | 1% Colloidal Oatmeal Eczema Cream | EpiCeram® Skin Barrier Emulsion
Number analyzed (Participants) | 39 | 12
participants
  I don't have an opinion | 0 | 0
  Strongly disagree | 1 | 1
  Somewhat disagree | 9 | 1
  Neither agree nor disagree | 3 | 1
  Somewhat agree | 15 | 6
  Strongly agree | 9 | 1
  Missing | 2 | 2

36. Secondary Outcome: Caregiver Questionnaire on Day 1 - Overall, my Baby's Skin Looks Healthy
Description: as for outcome 25
Time Frame: 1 Day
Population: Analysis was based on Intent-to-Treat subjects, which included all randomized subjects.
Measure: Number; unit: participants
Arm/Group | 1% Colloidal Oatmeal Eczema Cream | EpiCeram® Skin Barrier Emulsion
Number analyzed (Participants) | 39 | 12
participants
  I don't have an opinion | 0 | 0
  Strongly disagree | 1 | 1
  Somewhat disagree | 8 | 1
  Neither agree nor disagree | 5 | 0
  Somewhat agree | 16 | 7
  Strongly agree | 7 | 1
  Missing | 2 | 2

37. Secondary Outcome: Caregiver Questionnaire on Day 1 - Overall, my Baby's Skin Feels Soft
Description: as for outcome 25
Time Frame: 1 Day
Population: Analysis was based on Intent-to-Treat subjects, which included all randomized subjects.
Measure: Number; unit: participants
Arm/Group | 1% Colloidal Oatmeal Eczema Cream | EpiCeram® Skin Barrier Emulsion
Number analyzed (Participants) | 39 | 12
participants
  I don't have an opinion | 0 | 0
  Strongly disagree | 1 | 1
  Somewhat disagree | 10 | 1
  Neither agree nor disagree | 3 | 2
  Somewhat agree | 17 | 5
  Strongly agree | 6 | 1
  Missing | 2 | 2

38. Secondary Outcome: Caregiver Questionnaire on Day 1 - Overall, my Baby's Skin Feels Smooth
Description: as for outcome 25
Time Frame: 1 Day
Population: Analysis was based on Intent-to-Treat subjects, which included all randomized subjects.
Measure: Number; unit: participants
Arm/Group | 1% Colloidal Oatmeal Eczema Cream | EpiCeram® Skin Barrier Emulsion
Number analyzed (Participants) | 39 | 12
participants
  I don't have an opinion | 0 | 0
  Strongly disagree | 1 | 1
  Somewhat disagree | 9 | 1
  Neither agree nor disagree | 5 | 3
  Somewhat agree | 17 | 4
  Strongly agree | 5 | 1
  Missing | 2 | 2

39. Secondary Outcome: Caregiver Questionnaire on Day 1 - In the Areas Affected by Eczema, my Baby's Skin Looks Smooth
Description: as for outcome 25
Time Frame: 1 Day
Population: Analysis was based on Intent-to-Treat subjects, which included all randomized subjects.
Measure: Number; unit: participants
Arm/Group | 1% Colloidal Oatmeal Eczema Cream | EpiCeram® Skin Barrier Emulsion
Number analyzed (Participants) | 39 | 12
participants
  I don't have an opinion | 0 | 0
  Strongly disagree | 4 | 1
  Somewhat disagree | 13 | 5
  Neither agree nor disagree | 3 | 2
  Somewhat agree | 14 | 2
  Strongly agree | 3 | 0
  Missing | 2 | 2

40. Secondary Outcome: Caregiver Questionnaire on Day 1 - In the Areas Affected by Eczema, my Baby's Skin Looks Healthy
Description: as for outcome 25
Time Frame: 1 Day
Population: Analysis was based on Intent-to-Treat subjects, which included all randomized subjects.
Measure: Number; unit: participants
Arm/Group | 1% Colloidal Oatmeal Eczema Cream | EpiCeram® Skin Barrier Emulsion
Number analyzed (Participants) | 39 | 12
participants
  I don't have an opinion | 0 | 0
  Strongly disagree | 5 | 1
  Somewhat disagree | 11 | 6
  Neither agree nor disagree | 7 | 0
  Somewhat agree | 11 | 3
  Strongly agree | 3 | 0
  Missing | 2 | 2

41. Secondary Outcome: Caregiver Questionnaire on Day 1 - In the Areas Affected by Eczema, my Baby's Skin Feels Soft
Description: as for outcome 25
Time Frame: 1 Day
Population: Analysis was based on Intent-to-Treat subjects, which included all randomized subjects.
Measure: Number; unit: participants
Arm/Group | 1% Colloidal Oatmeal Eczema Cream | EpiCeram® Skin Barrier Emulsion
Number analyzed (Participants) | 39 | 12
participants
  I don't have an opinion | 0 | 0
  Strongly disagree | 4 | 1
  Somewhat disagree | 11 | 4
  Neither agree nor disagree | 1 | 1
  Somewhat agree | 16 | 4
  Strongly agree | 5 | 0
  Missing | 2 | 2

42. Secondary Outcome: Caregiver Questionnaire on Day 1 - In the Areas Affected by Eczema, my Baby's Skin Feels Smooth
Description: as for outcome 25
Time Frame: 1 Day
Population: Analysis was based on Intent-to-Treat subjects, which included all randomized subjects.
Measure: Number; unit: participants
Arm/Group | 1% Colloidal Oatmeal Eczema Cream | EpiCeram® Skin Barrier Emulsion
Number analyzed (Participants) | 39 | 12
participants
  I don't have an opinion | 0 | 0
  Strongly disagree | 5 | 1
  Somewhat disagree | 10 | 3
  Neither agree nor disagree | 4 | 2
  Somewhat agree | 13 | 4
  Strongly agree | 5 | 0
  Missing | 2 | 2

43. Secondary Outcome: Caregiver Questionnaire on Day 2 - Overall, my Baby's Skin Looks Smooth
Description: as for outcome 25
Time Frame: 2 Days
Population: Analysis was based on Intent-to-Treat subjects, which included all randomized subjects.
Measure: Number; unit: participants
Arm/Group | 1% Colloidal Oatmeal Eczema Cream | EpiCeram® Skin Barrier Emulsion
Number analyzed (Participants) | 39 | 12
participants
  I don't have an opinion | 0 | 0
  Strongly disagree | 1 | 1
  Somewhat disagree | 5 | 2
  Neither agree nor disagree | 2 | 0
  Somewhat agree | 16 | 6
  Strongly agree | 12 | 2
  Missing | 3 | 1

44. Secondary Outcome: Caregiver Questionnaire on Day 2 - Overall, my Baby's Skin Looks Healthy
Description: as for outcome 25
Time Frame: 2 Days
Population: Analysis was based on Intent-to-Treat subjects, which included all randomized subjects.
Measure: Number; unit: participants
Arm/Group | 1% Colloidal Oatmeal Eczema Cream | EpiCeram® Skin Barrier Emulsion
Number analyzed (Participants) | 39 | 12
participants
  I don't have an opinion | 0 | 0
  Strongly disagree | 1 | 1
  Somewhat disagree | 3 | 2
  Neither agree nor disagree | 5 | 1
  Somewhat agree | 18 | 5
  Strongly agree | 9 | 2
  Missing | 3 | 1

45. Secondary Outcome: Caregiver Questionnaire on Day 2 - Overall, my Baby's Skin Feels Soft
Description: as for outcome 25
Time Frame: 2 Days
Population: Analysis was based on Intent-to-Treat subjects, which included all randomized subjects.
Measure: Number; unit: participants
Arm/Group | 1% Colloidal Oatmeal Eczema Cream | EpiCeram® Skin Barrier Emulsion
Number analyzed (Participants) | 39 | 12
participants
  I don't have an opinion | 0 | 0
  Strongly disagree | 1 | 1
  Somewhat disagree | 4 | 1
  Neither agree nor disagree | 1 | 1
  Somewhat agree | 23 | 6
  Strongly agree | 7 | 2
  Missing | 3 | 1

46. Secondary Outcome: Caregiver Questionnaire on Day 2 - Overall, my Baby's Skin Feels Smooth
Description: as for outcome 25
Time Frame: 2 Days
Population: Analysis was based on Intent-to-Treat subjects, which included all randomized subjects.
Measure: Number; unit: participants
Arm/Group | 1% Colloidal Oatmeal Eczema Cream | EpiCeram® Skin Barrier Emulsion
Number analyzed (Participants) | 39 | 12
participants
  I don't have an opinion | 0 | 0
  Strongly disagree | 1 | 1
  Somewhat disagree | 6 | 2
  Neither agree nor disagree | 1 | 0
  Somewhat agree | 21 | 6
  Strongly agree | 7 | 2
  Missing | 3 | 1

47. Secondary Outcome: Caregiver Questionnaire on Day 2 - In the Areas Affected by Eczema, my Baby's Skin Looks Smooth
Description: as for outcome 25
Time Frame: 2 Days
Population: Analysis was based on Intent-to-Treat subjects, which included all randomized subjects.
Measure: Number; unit: participants
Arm/Group | 1% Colloidal Oatmeal Eczema Cream | EpiCeram® Skin Barrier Emulsion
Number analyzed (Participants) | 39 | 12
participants
  I don't have an opinion | 0 | 0
  Strongly disagree | 3 | 2
  Somewhat disagree | 9 | 3
  Neither agree nor disagree | 1 | 1
  Somewhat agree | 17 | 4
  Strongly agree | 6 | 1
  Missing | 3 | 1

48. Secondary Outcome: Caregiver Questionnaire on Day 2 - In the Areas Affected by Eczema, my Baby's Skin Looks Healthy
Description: as for outcome 25
Time Frame: 2 Days
Population: Analysis was based on Intent-to-Treat subjects, which included all randomized subjects.
Measure: Number; unit: participants
Arm/Group | 1% Colloidal Oatmeal Eczema Cream | EpiCeram® Skin Barrier Emulsion
Number analyzed (Participants) | 39 | 12
participants
  I don't have an opinion | 0 | 0
  Strongly disagree | 3 | 2
  Somewhat disagree | 8 | 4
  Neither agree nor disagree | 5 | 0
  Somewhat agree | 16 | 4
  Strongly agree | 4 | 1
  Missing | 3 | 1

49. Secondary Outcome: Caregiver Questionnaire on Day 2 - In the Areas Affected by Eczema, my Baby's Skin Feels Soft
Description: as for outcome 25
Time Frame: 2 Days
Population: Analysis was based on Intent-to-Treat subjects, which included all randomized subjects.
Measure: Number; unit: participants
Arm/Group | 1% Colloidal Oatmeal Eczema Cream | EpiCeram® Skin Barrier Emulsion
Number analyzed (Participants) | 39 | 12
participants
  I don't have an opinion | 0 | 0
  Strongly disagree | 2 | 2
  Somewhat disagree | 10 | 2
  Neither agree nor disagree | 4 | 1
  Somewhat agree | 13 | 5
  Strongly agree | 7 | 1
  Missing | 3 | 1

50. Secondary Outcome: Caregiver Questionnaire on Day 2 - In the Areas Affected by Eczema, my Baby's Skin Feels Smooth
Description: as for outcome 25
Time Frame: 2 Days
Population: Analysis was based on Intent-to-Treat subjects, which included all randomized subjects.
Measure: Number; unit: participants
Arm/Group | 1% Colloidal Oatmeal Eczema Cream | EpiCeram® Skin Barrier Emulsion
Number analyzed (Participants) | 39 | 12
participants
  I don't have an opinion | 0 | 0
  Strongly disagree | 3 | 2
  Somewhat disagree | 13 | 2
  Neither agree nor disagree | 0 | 1
  Somewhat agree | 13 | 5
  Strongly agree | 7 | 1
  Missing | 3 | 1

51. Secondary Outcome: Caregiver Questionnaire on Day 3 - Overall, my Baby's Skin Looks Smooth
Description: as for outcome 25
Time Frame: 3 Days
Population: Analysis was based on Intent-to-Treat subjects, which included all randomized subjects.
Measure: Number; unit: participants
Arm/Group | 1% Colloidal Oatmeal Eczema Cream | EpiCeram® Skin Barrier Emulsion
Number analyzed (Participants) | 39 | 12
participants
  I don't have an opinion | 0 | 0
  Strongly disagree | 1 | 1
  Somewhat disagree | 2 | 1
  Neither agree nor disagree | 3 | 1
  Somewhat agree | 19 | 5
  Strongly agree | 9 | 3
  Missing | 5 | 1

52. Secondary Outcome: Caregiver Questionnaire on Day 3 - Overall, my Baby's Skin Looks Healthy
Description: as for outcome 25
Time Frame: 3 Days
Population: Analysis was based on Intent-to-Treat subjects, which included all randomized subjects.
Measure: Number; unit: participants
Arm/Group | 1% Colloidal Oatmeal Eczema Cream | EpiCeram® Skin Barrier Emulsion
Number analyzed (Participants) | 39 | 12
participants
  I don't have an opinion | 0 | 0
  Strongly disagree | 1 | 1
  Somewhat disagree | 3 | 1
  Neither agree nor disagree | 5 | 1
  Somewhat agree | 18 | 5
  Strongly agree | 7 | 3
  Missing | 5 | 1

53. Secondary Outcome: Caregiver Questionnaire on Day 3 - Overall, my Baby's Skin Feels Soft
Description: as for outcome 25
Time Frame: 3 Days
Population: Analysis was based on Intent-to-Treat subjects, which included all randomized subjects.
Measure: Number; unit: participants
Arm/Group | 1% Colloidal Oatmeal Eczema Cream | EpiCeram® Skin Barrier Emulsion
Number analyzed (Participants) | 39 | 12
participants
  I don't have an opinion | 0 | 0
  Strongly disagree | 1 | 1
  Somewhat disagree | 6 | 0
  Neither agree nor disagree | 1 | 1
  Somewhat agree | 18 | 6
  Strongly agree | 8 | 3
  Missing | 5 | 1

54. Secondary Outcome: Caregiver Questionnaire on Day 3 - Overall, my Baby's Skin Feels Smooth
Description: as for outcome 25
Time Frame: 3 Days
Population: Analysis was based on Intent-to-Treat subjects, which included all randomized subjects.
Measure: Number; unit: participants
Arm/Group | 1% Colloidal Oatmeal Eczema Cream | EpiCeram® Skin Barrier Emulsion
Number analyzed (Participants) | 39 | 12
participants
  I don't have an opinion | 0 | 0
  Strongly disagree | 1 | 1
  Somewhat disagree | 5 | 1
  Neither agree nor disagree | 1 | 1
  Somewhat agree | 19 | 5
  Strongly agree | 8 | 3
  Missing | 5 | 1

55. Secondary Outcome: Caregiver Questionnaire on Day 3 - In the Areas Affected by Eczema, my Baby's Skin Looks Smooth
Description: as for outcome 25
Time Frame: 3 Days
Population: Analysis was based on Intent-to-Treat subjects, which included all randomized subjects.
Measure: Number; unit: participants
Arm/Group | 1% Colloidal Oatmeal Eczema Cream | EpiCeram® Skin Barrier Emulsion
Number analyzed (Participants) | 39 | 12
participants
  I don't have an opinion | 0 | 0
  Strongly disagree | 2 | 1
  Somewhat disagree | 8 | 2
  Neither agree nor disagree | 2 | 1
  Somewhat agree | 15 | 5
  Strongly agree | 7 | 2
  Missing | 5 | 1

56. Secondary Outcome: Caregiver Questionnaire on Day 3 - In the Areas Affected by Eczema, my Baby's Skin Looks Healthy
Description: as for outcome 25
Time Frame: 3 Days
Population: Analysis was based on Intent-to-Treat subjects, which included all randomized subjects.
Measure: Number; unit: participants
Arm/Group | 1% Colloidal Oatmeal Eczema Cream | EpiCeram® Skin Barrier Emulsion
Number analyzed (Participants) | 39 | 12
participants
  I don't have an opinion | 0 | 0
  Strongly disagree | 2 | 1
  Somewhat disagree | 7 | 2
  Neither agree nor disagree | 4 | 2
  Somewhat agree | 16 | 5
  Strongly agree | 5 | 1
  Missing | 5 | 1

57. Secondary Outcome: Caregiver Questionnaire on Day 3 - In the Areas Affected by Eczema, my Baby's Skin Feels Soft
Description: as for outcome 25
Time Frame: 3 Days
Population: Analysis was based on Intent-to-Treat subjects, which included all randomized subjects.
Measure: Number; unit: participants
Arm/Group | 1% Colloidal Oatmeal Eczema Cream | EpiCeram® Skin Barrier Emulsion
Number analyzed (Participants) | 39 | 12
participants
  I don't have an opinion | 0 | 0
  Strongly disagree | 2 | 1
  Somewhat disagree | 8 | 3
  Neither agree nor disagree | 4 | 1
  Somewhat agree | 10 | 5
  Strongly agree | 10 | 1
  Missing | 5 | 1

58. Secondary Outcome: Caregiver Questionnaire on Day 3 - In the Areas Affected by Eczema, my Baby's Skin Feels Smooth
Description: as for outcome 25
Time Frame: 3 Days
Population: Analysis was based on Intent-to-Treat subjects, which included all randomized subjects.
Measure: Number; unit: participants
Arm/Group | 1% Colloidal Oatmeal Eczema Cream | EpiCeram® Skin Barrier Emulsion
Number analyzed (Participants) | 39 | 12
participants
  I don't have an opinion | 0 | 0
  Strongly disagree | 2 | 1
  Somewhat disagree | 9 | 3
  Neither agree nor disagree | 2 | 1
  Somewhat agree | 12 | 5
  Strongly agree | 9 | 1
  Missing | 5 | 1

59. Secondary Outcome: Caregiver Questionnaire on Day 7 - Overall, my Baby's Skin Looks Smooth
Description: as for outcome 25
Time Frame: 7 Days
Population: Analysis was based on Intent-to-Treat subjects, which included all randomized subjects.
Measure: Number; unit: participants
Arm/Group | 1% Colloidal Oatmeal Eczema Cream | EpiCeram® Skin Barrier Emulsion
Number analyzed (Participants) | 39 | 12
participants
  I don't have an opinion | 0 | 0
  Strongly disagree | 2 | 1
  Somewhat disagree | 1 | 1
  Neither agree nor disagree | 2 | 0
  Somewhat agree | 13 | 5
  Strongly agree | 17 | 4
  Missing | 4 | 1

60. Secondary Outcome: Caregiver Questionnaire on Day 7 - Overall, my Baby's Skin Looks Healthy
Description: as for outcome 25
Time Frame: 7 Days
Population: Analysis was based on Intent-to-Treat subjects, which included all randomized subjects.
Measure: Number; unit: participants
Arm/Group | 1% Colloidal Oatmeal Eczema Cream | EpiCeram® Skin Barrier Emulsion
Number analyzed (Participants) | 39 | 12
participants
  I don't have an opinion | 0 | 0
  Strongly disagree | 2 | 1
  Somewhat disagree | 1 | 1
  Neither agree nor disagree | 3 | 1
  Somewhat agree | 15 | 3
  Strongly agree | 14 | 5
  Missing | 4 | 1

61. Secondary Outcome: Caregiver Questionnaire on Day 7 - Overall, my Baby's Skin Feels Soft
Description: as for outcome 25
Time Frame: 7 Days
Population: Analysis was based on Intent-to-Treat subjects, which included all randomized subjects.
Measure: Number; unit: participants
Arm/Group | 1% Colloidal Oatmeal Eczema Cream | EpiCeram® Skin Barrier Emulsion
Number analyzed (Participants) | 39 | 12
participants
  I don't have an opinion | 0 | 0
  Strongly disagree | 2 | 1
  Somewhat disagree | 0 | 2
  Neither agree nor disagree | 3 | 0
  Somewhat agree | 16 | 4
  Strongly agree | 14 | 4
  Missing | 4 | 1

62. Secondary Outcome: Caregiver Questionnaire on Day 7 - Overall, my Baby's Skin Feels Smooth
Description: as for outcome 25
Time Frame: 7 Days
Population: Analysis was based on Intent-to-Treat subjects, which included all randomized subjects.
Measure: Number; unit: participants
Arm/Group | 1% Colloidal Oatmeal Eczema Cream | EpiCeram® Skin Barrier Emulsion
Number analyzed (Participants) | 39 | 12
participants
  I don't have an opinion | 0 | 0
  Strongly disagree | 2 | 1
  Somewhat disagree | 2 | 2
  Neither agree nor disagree | 1 | 0
  Somewhat agree | 19 | 4
  Strongly agree | 11 | 4
  Missing | 4 | 1

63. Secondary Outcome: Caregiver Questionnaire on Day 7 - In the Areas Affected by Eczema, my Baby's Skin Looks Smooth
Description: as for outcome 25
Time Frame: 7 Days
Population: Analysis was based on Intent-to-Treat subjects, which included all randomized subjects.
Measure: Number; unit: participants
Arm/Group | 1% Colloidal Oatmeal Eczema Cream | EpiCeram® Skin Barrier Emulsion
Number analyzed (Participants) | 39 | 12
participants
  I don't have an opinion | 0 | 0
  Strongly disagree | 2 | 1
  Somewhat disagree | 5 | 2
  Neither agree nor disagree | 2 | 2
  Somewhat agree | 12 | 3
  Strongly agree | 14 | 3
  Missing | 4 | 1

64. Secondary Outcome: Caregiver Questionnaire on Day 7 - In the Areas Affected by Eczema, my Baby's Skin Looks Healthy
Description: as for outcome 25
Time Frame: 7 Days
Population: Analysis was based on Intent-to-Treat subjects, which included all randomized subjects.
Measure: Number; unit: participants
Arm/Group | 1% Colloidal Oatmeal Eczema Cream | EpiCeram® Skin Barrier Emulsion
Number analyzed (Participants) | 39 | 12
participants
  I don't have an opinion | 0 | 0
  Strongly disagree | 2 | 1
  Somewhat disagree | 4 | 3
  Neither agree nor disagree | 2 | 1
  Somewhat agree | 16 | 3
  Strongly agree | 11 | 3
  Missing | 4 | 1

65. Secondary Outcome: Caregiver Questionnaire on Day 7 - In the Areas Affected by Eczema, my Baby's Skin Feels Soft
Description: as for outcome 25
Time Frame: 7 Days
Population: Analysis was based on Intent-to-Treat subjects, which included all randomized subjects.
Measure: Number; unit: participants
Arm/Group | 1% Colloidal Oatmeal Eczema Cream | EpiCeram® Skin Barrier Emulsion
Number analyzed (Participants) | 39 | 12
participants
  I don't have an opinion | 0 | 0
  Strongly disagree | 2 | 1
  Somewhat disagree | 4 | 2
  Neither agree nor disagree | 6 | 1
  Somewhat agree | 7 | 4
  Strongly agree | 16 | 3
  Missing | 4 | 1

66. Secondary Outcome: Caregiver Questionnaire on Day 7 - In the Areas Affected by Eczema, my Baby's Skin Feels Smooth
Description: as for outcome 25
Time Frame: 7 Days
Population: Analysis was based on Intent-to-Treat subjects, which included all randomized subjects.
Measure: Number; unit: participants
Arm/Group | 1% Colloidal Oatmeal Eczema Cream | EpiCeram® Skin Barrier Emulsion
Number analyzed (Participants) | 39 | 12
participants
  I don't have an opinion | 0 | 0
  Strongly disagree | 2 | 1
  Somewhat disagree | 5 | 2
  Neither agree nor disagree | 5 | 2
  Somewhat agree | 11 | 3
  Strongly agree | 12 | 3
  Missing | 4 | 1

67. Secondary Outcome: Caregiver Questionnaire on Day 14 - Overall, my Baby's Skin Looks Smooth
Description: as for outcome 25
Time Frame: 14 Days
Population: Analysis was based on Intent-to-Treat subjects, which included all randomized subjects.
Measure: Number; unit: participants
Arm/Group | 1% Colloidal Oatmeal Eczema Cream | EpiCeram® Skin Barrier Emulsion
Number analyzed (Participants) | 39 | 12
participants
  I don't have an opinion | 0 | 0
  Strongly disagree | 1 | 1
  Somewhat disagree | 3 | 0
  Neither agree nor disagree | 2 | 0
  Somewhat agree | 11 | 3
  Strongly agree | 19 | 7
  Missing | 3 | 1

68. Secondary Outcome: Caregiver Questionnaire on Day 14 - Overall, my Baby's Skin Looks Healthy
Description: as for outcome 25
Time Frame: 14 Days
Population: Analysis was based on Intent-to-Treat subjects, which included all randomized subjects.
Measure: Number; unit: participants
Arm/Group | 1% Colloidal Oatmeal Eczema Cream | EpiCeram® Skin Barrier Emulsion
Number analyzed (Participants) | 39 | 12
participants
  I don't have an opinion | 0 | 0
  Strongly disagree | 1 | 1
  Somewhat disagree | 3 | 0
  Neither agree nor disagree | 1 | 0
  Somewhat agree | 14 | 4
  Strongly agree | 17 | 6
  Missing | 3 | 1

69. Secondary Outcome: Caregiver Questionnaire on Day 14 - Overall, my Baby's Skin Feels Soft
Description: as for outcome 25
Time Frame: 14 Days
Population: Analysis was based on Intent-to-Treat subjects, which included all randomized subjects.
Measure: Number; unit: participants
Arm/Group | 1% Colloidal Oatmeal Eczema Cream | EpiCeram® Skin Barrier Emulsion
Number analyzed (Participants) | 39 | 12
participants
  I don't have an opinion | 0 | 0
  Strongly disagree | 1 | 1
  Somewhat disagree | 1 | 0
  Neither agree nor disagree | 4 | 0
  Somewhat agree | 15 | 3
  Strongly agree | 15 | 7
  Missing | 3 | 1

70. Secondary Outcome: Caregiver Questionnaire on Day 14 - Overall, my Baby's Skin Feels Smooth
Description: as for outcome 25
Time Frame: 14 Days
Population: Analysis was based on Intent-to-Treat subjects, which included all randomized subjects.
Measure: Number; unit: participants
Arm/Group | 1% Colloidal Oatmeal Eczema Cream | EpiCeram® Skin Barrier Emulsion
Number analyzed (Participants) | 39 | 12
participants
  I don't have an opinion | 0 | 0
  Strongly disagree | 1 | 1
  Somewhat disagree | 2 | 0
  Neither agree nor disagree | 3 | 0
  Somewhat agree | 13 | 3
  Strongly agree | 17 | 7
  Missing | 3 | 1

71. Secondary Outcome: Caregiver Questionnaire on Day 14 - In the Areas Affected by Eczema, my Baby's Skin Looks Smooth
Description: as for outcome 25
Time Frame: 14 Days
Population: Analysis was based on Intent-to-Treat subjects, which included all randomized subjects.
Measure: Number; unit: participants
Arm/Group | 1% Colloidal Oatmeal Eczema Cream | EpiCeram® Skin Barrier Emulsion
Number analyzed (Participants) | 39 | 12
participants
  I don't have an opinion | 0 | 0
  Strongly disagree | 2 | 1
  Somewhat disagree | 1 | 0
  Neither agree nor disagree | 3 | 2
  Somewhat agree | 13 | 4
  Strongly agree | 17 | 4
  Missing | 3 | 1

72. Secondary Outcome: Caregiver Questionnaire on Day 14 - In the Areas Affected by Eczema, my Baby's Skin Looks Healthy
Description: as for outcome 25
Time Frame: 14 Days
Population: Analysis was based on Intent-to-Treat subjects, which included all randomized subjects.
Measure: Number; unit: participants
Arm/Group | 1% Colloidal Oatmeal Eczema Cream | EpiCeram® Skin Barrier Emulsion
Number analyzed (Participants) | 39 | 12
participants
  I don't have an opinion | 0 | 0
  Strongly disagree | 2 | 1
  Somewhat disagree | 0 | 1
  Neither agree nor disagree | 3 | 1
  Somewhat agree | 14 | 4
  Strongly agree | 17 | 4
  Missing | 3 | 1

73. Secondary Outcome: Caregiver Questionnaire on Day 14 - In the Areas Affected by Eczema, my Baby's Skin Feels Soft
Description: as for outcome 25
Time Frame: 14 Days
Population: Analysis was based on Intent-to-Treat subjects, which included all randomized subjects.
Measure: Number; unit: participants
Arm/Group | 1% Colloidal Oatmeal Eczema Cream | EpiCeram® Skin Barrier Emulsion
Number analyzed (Participants) | 39 | 12
participants
  I don't have an opinion | 0 | 0
  Strongly disagree | 2 | 1
  Somewhat disagree | 1 | 0
  Neither agree nor disagree | 2 | 0
  Somewhat agree | 14 | 6
  Strongly agree | 17 | 4
  Missing | 3 | 1

74. Secondary Outcome: Caregiver Questionnaire on Day 14 - In the Areas Affected by Eczema, my Baby's Skin Feels Smooth
Description: as for outcome 25
Time Frame: 14 Days
Population: Analysis was based on Intent-to-Treat subjects, which included all randomized subjects.
Measure: Number; unit: participants
Arm/Group | 1% Colloidal Oatmeal Eczema Cream | EpiCeram® Skin Barrier Emulsion
Number analyzed (Participants) | 39 | 12
participants
  I don't have an opinion | 0 | 0
  Strongly disagree | 2 | 1
  Somewhat disagree | 1 | 0
  Neither agree nor disagree | 2 | 0
  Somewhat agree | 11 | 6
  Strongly agree | 20 | 4
  Missing | 3 | 1

75. Secondary Outcome: Caregiver Questionnaire on Day 14 - I Would Recommend This Product to Another Parent.
Description: Questions were answered immediately post-treatment by participant's caregiver. Caregiver answered based on a 6 point system from 'I don't have an opinion' to 'strongly disagree.'
Time Frame: 14 Days
Population: Analysis was based on Intent-to-Treat subjects, which included all randomized subjects.
Measure: Number; unit: participants
Arm/Group | 1% Colloidal Oatmeal Eczema Cream | EpiCeram® Skin Barrier Emulsion
Number analyzed (Participants) | 39 | 12
participants
  I don't have an opinion | 1 | 0
  Strongly disagree | 1 | 1
  Somewhat disagree | 0 | 0
  Neither agree nor disagree | 2 | 1
  Somewhat agree | 9 | 1
  Strongly agree | 23 | 8
  Missing | 3 | 1

ADVERSE EVENTS:
Time Frame: Day 14 ± 1 day, +30 days for serious adverse events.
Description: Adverse events were systematically collected at each study visit through Visit 6 (Day 14 ± 1 day). Serious adverse events were reported through 30 days after product use. Spontaneously reported adverse events collected outside of the regularly scheduled visits were also recorded.
Arm/Group | 1% Colloidal Oatmeal Eczema Cream | EpiCeram® Skin Barrier Emulsion
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/12
Other Adverse Events (participants affected / at risk) | 0/39 | 1/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 1% Colloidal Oatmeal Eczema Cream (N=39) | EpiCeram® Skin Barrier Emulsion (N=12)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal investigator agreed not to publish the study results without prior sponsor approval.